CLINICAL TRIAL: NCT04903925
Title: Efficacy of Probiotics in Improving Post-surgical Healing for Impacted Tooth Extractions
Brief Title: Probiotics for Improving Post-surgical Healing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Antonio Barone, Professor, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Antib Prob Impacted 1
Record Dates: First submitted 2021-05-18; First posted 2021-05-27 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Probiotics; Tooth, Impacted; Wound Heal; Gastrointestinal Complication
MeSH Terms: conditions — Tooth, Impacted

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): All patients will undergo an impacted tooth extraction; patients allocated to group 1 will receive an antibiotic therapy with amoxicillin for 6 days (2 g/day) and a probiotic for 21 days (2 tablets/day).
  Interventions: Procedure: Impacted tooth extraction
- Group 2 (Placebo Comparator): All patients will undergo an impacted tooth extraction; patients allocated to group 1 will receive an antibiotic therapy with amoxicillin for 6 days (2 g/day) and a placebo of the probiotic for 21 days (2 tablets/day).
  Interventions: Procedure: Impacted tooth extraction

INTERVENTIONS:
Procedure: Impacted tooth extraction — All patients will undergo a surgical tooth extraction

SUMMARY:
A randomized, double-blind, placebo-controlled clinical trial will be performed to assess the efficacy of a probiotic containing Lactobacillus reuteri in improving post-surgical wound healing after impacted tooth extractions.

The Primary aim is to evaluate the efficacy of L. reuteri in improving post-extractive healing.

The Secondary aim is to evaluate the efficacy of L. reuteri in association with an antibiotic therapy (amoxicillin) in reducing the incidence and severity of antibiotic-associated gastro-intestinal symptoms.

DETAILED DESCRIPTION:
Probiotics are defined by the World Health Organization as "live microorganisms which, when administered in adequate amounts, confer a health benefit on the host." Human microbiome is a complex system that contributes to maintaining a good health status in humans. Broad-spectrum antibiotic therapies act against pathogen bacteria but also affect the intestinal microbiome, leading to different side effects such as abdominal pain, gastric pain, nausea, vomit and diarrhea.

The use of probiotics has been advocated as a possible means in reducing intensity and incidence of the symptoms related to antibiotic therapies. Some probiotics like Lactobacillus reuteri (L. reuteri) showed good anti-inflammatory properties and also antimicrobic action, assuming a possible role in wound healing processes.

Few studies have been conducted on the use of L. reuteri in dentistry. Twetman et al. (2018) conducted a trial to assess the efficacy of L. reuteri in improving post-surgical healing in the oral cavity after a punch biopsy, showing promising results. The authors concluded that larger trials may be useful to better clarify the role of probiotics in oral wounds healing. The only data regarding the possible role of L. reuteri in post- extractive healing comes from a pilot study (Walivara at al. 2019) that showed a reduction of the perceived swelling and of the number of disturbed-sleep nights in patients who underwent impacted-tooth extraction and assumed L. reuteri. Authors concluded that larger trials with closer follow-up visits are required to fully understand the clinical correlation.

The primary aim of the present research is to evaluate the efficacy of a probiotic containing L. reuteri in improving post-surgical healing following impacted tooth extractions and the secondary aim is to investigate its possible role in preventing or reducing gastro-intestinal side effects related to post-operative antibiotic therapy.A Randomized, double-blind, placebo-controlled clinical trial will be performed to evaluate the efficacy of L. reuteri in improving post-extractive healing.

All patients who need impacted tooth extractions at University Hospital of Pisa (Operative Unit of Odontostomatology and Oral Surgery) will be considered eligible for the study.

The number of patients to include is set to 160, divided in two experimental groups (80 patients per group). Patients who meet inclusion/exclusion criteria will be enrolled in this trial.

ELIGIBILITY:
Inclusion Criteria:

* need for impacted tooth extractions
* over age 18
* ability to understand and to sign an informed consent form

Exclusion Criteria:

* allergy to penicillin
* contraindications to oral surgery
* treatment with immunosuppressive agents or immunocompromised
* treatment with amino-bisphosphonate and anti-angiogenetic medications
* irradiation to head and neck area
* uncontrolled diabetes
* renal failure
* drug and alcohol addiction
* psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-04-13 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Surgical wound healing | 3 days after the surgery
  Clinical assessment of the characteristics of the surgical wound
Surgical wound healing | 7 days after the surgery
  Clinical assessment of the characteristics of the surgical wound
Surgical wound healing | 14 days after the surgery
  Clinical assessment of the characteristics of the surgical wound

SECONDARY OUTCOMES:
Presence of pain | 3 days after the surgery
  presence of pain assessed by VAS (0-10)
Presence of pain | 7 days after the surgery
  presence of pain assessed by VAS (0-10)
Presence of pain | 14 days after the surgery
  presence of pain assessed by VAS (0-10)
Abscess | 3 days after the surgery
  presence of suppuration
Abscess | 7 days after the surgery
  presence of suppuration
Abscess | 14 days after the surgery
  presence of suppuration
Edema | 3 days after the surgery
  presence and evaluation of the post-operative edema (intra-oral and extra-oral)
Edema | 7 days after the surgery
  presence and evaluation of the post-operative edema (intra-oral and extra-oral)
Edema | 14 days after the surgery
  presence and evaluation of the post-operative edema (intra-oral and extra-oral)
Fever | 3 days after the surgery
  Body temperature > 37°C
Fever | 7 days after the surgery
  Body temperature > 37°C
Fever | 14 days after the surgery
  Body temperature > 37°C
Alveolar osteitis | 3 days after the surgery
  Presence of alveolar osteitis
Alveolar osteitis | 7 days after the surgery
  Presence of alveolar osteitis
Alveolar osteitis | 14 days after the surgery
  Presence of alveolar osteitis
Trismus | 3 days after the surgery
  reduction in mouth opening (measured in mm)
Trismus | 7 days after the surgery
  reduction in mouth opening (measured in mm)
Trismus | 14 days after the surgery
  reduction in mouth opening (measured in mm)
Painkillers | 7 days after the surgery
  Number of painkillers assumed in the first 7 days after the surgery
bleeding on palpation | 3 days after the surgery
  presence of bleeding on palpation
bleeding on palpation | 7 days after the surgery
  presence of bleeding on palpation
bleeding on palpation | 14 days after the surgery
  presence of bleeding on palpation
Difficulty in chewing | 3 days after the surgery
  Difficulty in chewing assessed by VAS (0-10)
Difficulty in chewing | 7 days after the surgery
  Difficulty in chewing assessed by VAS (0-10)
Difficulty in chewing | 14 days after the surgery
  Difficulty in chewing assessed by VAS (0-10)
Difficulty in speaking | 3 days after the surgery
  Difficulty in speaking assessed by VAS (0-10)
Difficulty in speaking | 7 days after the surgery
  Difficulty in speaking assessed by VAS (0-10)
Difficulty in speaking | 14 days after the surgery
  Difficulty in speaking assessed by VAS (0-10)
Difficulty in performing oral hygiene | 3 days after the surgery
  Difficulty in performing oral hygiene assessed by VAS (0-10)
Difficulty in performing oral hygiene | 7 days after the surgery
  Difficulty in performing oral hygiene assessed by VAS (0-10)
Difficulty in performing oral hygiene | 14 days after the surgery
  Difficulty in performing oral hygiene assessed by VAS (0-10)
Daily routine alterations | 3 days after the surgery
  days of stay off work
Daily routine alterations | 7 days after the surgery
  days of stay off work
Daily routine alterations | 14 days after the surgery
  days of stay off work
Sensation of swelling | 3 days after the surgery
  assessed by VAS (0-10)
Sensation of swelling | 7 days after the surgery
  assessed by VAS (0-10)
Sensation of swelling | 14 days after the surgery
  assessed by VAS (0-10)
Number of disturbed-sleep nights following the extraction | 3 days after the surgery
  Number of disturbed-sleep nights
Number of disturbed-sleep nights following the extraction | 7 days after the surgery
  Number of disturbed-sleep nights
Number of disturbed-sleep nights following the extraction | 14 days after the surgery
  Number of disturbed-sleep nights
Abdominal pain | 3 days after the surgery
  presence of Abdominal pain (questionnarie Y/N)
Abdominal pain | 7 days after the surgery
  presence of Abdominal pain (questionnarie Y/N)
Abdominal pain | 14 days after the surgery
  presence of Abdominal pain (questionnarie Y/N)
Abdominal distension | 3 days after the surgery
  presence of Abdominal pain (questionnarie Y/N)
Abdominal distension | 7 days after the surgery
  presence of Abdominal pain (questionnarie Y/N)
Abdominal distension | 14 days after the surgery
  presence of Abdominal pain (questionnarie Y/N)
Alvus variation | 3 days after the surgery
  presence of alvus variations (questionnarie Y/N)
Alvus variation | 7 days after the surgery
  presence of alvus variations (questionnarie Y/N)
Alvus variation | 14 days after the surgery
  presence of alvus variations (questionnarie Y/N)
Nausea | 3 days after the surgery
  presence of nausea (questionnarie Y/N)
Nausea | 7 days after the surgery
  presence of nausea (questionnarie Y/N)
Nausea | 14 days after the surgery
  presence of nausea (questionnarie Y/N)
Vomit | 3 days after the surgery
  presence of vomit (questionnarie Y/N)
Vomit | 7 days after the surgery
  presence of vomit (questionnarie Y/N)
Vomit | 14 days after the surgery
  presence of vomit (questionnarie Y/N)
Acid reflux | 3 days after the surgery
  presence of acid reflux (questionnarie Y/N)
Acid reflux | 7 days after the surgery
  presence of acid reflux (questionnarie Y/N)
Acid reflux | 14 days after the surgery
  presence of acid reflux (questionnarie Y/N)
Gastric acidity | 3 days after the surgery
  presence of gastric acidity (questionnarie Y/N)
Gastric acidity | 7 days after the surgery
  presence of gastric acidity (questionnarie Y/N)
Gastric acidity | 14 days after the surgery
  presence of gastric acidity (questionnarie Y/N)
Gastric pain | 3 days after the surgery
  presence of gastric pain (questionnarie Y/N)
Gastric pain | 7 days after the surgery
  presence of gastric pain (questionnarie Y/N)
Gastric pain | 14 days after the surgery
  presence of gastric pain (questionnarie Y/N)
Loss of appetite | 3 days after the surgery
  presence of loss of appetite (questionnarie Y/N)
Loss of appetite | 7 days after the surgery
  presence of loss of appetite (questionnarie Y/N)
Loss of appetite | 14 days after the surgery
  presence of loss of appetite (questionnarie Y/N)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Barone, Professor, Principal Investigator — University of Pisa
Locations (1):
- U.O. Odontostomatologia e Chirurgia del Cavo Orale, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cinquini C, Izzetti R, Nisi M, Gulia F, Garcia Mira B, Barone A. Limosilactobacillus reuteri Improves Healing Following Fully Impacted Tooth Extractions: Randomized Clinical Trial. Oral Dis. 2025 Jul 13. doi: 10.1111/odi.70026. Online ahead of print. PMID 40652540